CLINICAL TRIAL: NCT02171754
Title: Relative Bioavailability of a Single Oral Dose of BIBW 2992 (20 mg) After Coadministration With Multiple Oral Doses of Ritonavir (200 mg Bid for 3 Days) Compared to the Bioavailability of a Single Oral Dose of BIBW 2992 (20 mg) Alone in Healthy Male Volunteers (an Open-label, Randomised, Two-way Crossover, Clinical Phase I Study)
Brief Title: Relative Bioavailability of a Single-dose Administration of BIBW 2992 and Multiple-dose Administration of Ritonavir in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1200.79
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
MeSH Terms: interventions — Afatinib; Ritonavir

ARMS (2):
- BIBW 2992 + Ritonavir (Experimental)
  Interventions: Drug: BIBW 2992; Drug: Ritonavir
- BIBW 2992 (Active Comparator)
  Interventions: Drug: BIBW 2992

INTERVENTIONS:
Drug: BIBW 2992
Drug: Ritonavir
  Arms: BIBW 2992 + Ritonavir

SUMMARY:
The objective was to investigate the effect of ritonavir, an inhibitor of P-glycoprotein (P-gp) and cytochrome P450 3A4 (CYP3A4), on the pharmacokinetics of BIBW 2992

ELIGIBILITY:
Inclusion Criteria:

* Healthy males according to a complete medical history, including a physical examination, vital signs (blood pressure, pulse rate), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age 21 to 55 years, inclusive
* Body mass index 18.5 to 29.9 kg/m2, inclusive
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including Blood Pressure (BP), Pulse Rate (PR) and Electrocardiogram (ECG)) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts 7. Chronic or relevant acute infections (e.g. HIV)
* History of relevant allergy/hypersensitivity (including drug allergy or its excipients)
* Intake of drugs with a long half-life (>24 hours) within 1 month prior to administration of the trial drug or during the trial
* Use of any drugs (including herbal preparations, vitamins and nutrient supplements) within 14 days prior to first administration of the trial drug or during the trial
* Participation in another trial with an investigational drug within 2 months prior to administration or during the trial
* Smoker (>10 cigarettes or >3 cigars or >3 pipes/day)
* Inability to refrain from smoking within the in-house periods from 12 hours before until 25 hours after each administration of the trial drug
* Alcohol abuse (more than 30 g/day)
* Drug abuse
* Blood donation (more than 100 mL within 4 weeks prior to administration of the trial drug or during the trial)
* Excessive physical activities (within 1 week prior to administration of the trial drug or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (e.g. repeated demonstration of a QTc interval >450 ms)
* A history of additional risk factors for Torsades de Points, e.g. heart failure, hypokalemia, family history of Long QT Syndrome

Exclusion criteria specific for this study:

* History of clinically relevant skin diseases, psoriasis or moderate/severe acne
* History or evidence of interstitial lung disease
* Males who are unwilling to use a medically acceptable method of contraception during the first 3 months after administration of BIBW 2992. Acceptable methods of contraception for use by male volunteers include sexual abstinence, a vasectomy performed at least 1 year prior to dosing, barrier contraception or another medically accepted contraceptive method

Ages: 21 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2009-09; Primary Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to infinity) - BIBW 2992 | up to 6 days after drug administration
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point) - BIBW2992 | up to 6 days after drug administration
Cmax (maximum measured concentration of the analyte in plasma) - BIBW 2992 | up to 6 days after drug administration

SECONDARY OUTCOMES:
AUC0-24 (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to 24 hours) - BIBW 2992 | up to 6 days after drug administration
%AUCtz-∞ (percentage of the AUCtz-∞ that is obtained by extrapolation from the last quantifiable data point to infinity) - BIBW 2992 | up to 6 days after drug administration
tmax (time from dosing to the maximum concentration of the analyte in plasma) - BIBW 2992 | up to 6 days after drug administration
λz (terminal rate constant in plasma) - BIBW 2992 | up to 6 days after drug administration
t1/2 (terminal half-life of the analyte in plasma) - BIBW 2992 | up to 6 days after drug administration
MRTpo (mean residence time of the analyte in the body after oral administration) - BIBW 2992 | up to 6 days after drug administration
CL/F (apparent clearance of the analyte in the plasma after extravascular administration) - BIBW 2992 | up to 6 days after drug administration
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) - BIBW 2992 | up to 6 days after drug administration
Number of patients with abnormal findings in physical examination | Screening, up to 20 days after drug administration
Number of patients with clinically significant changes in vital signs (blood pressure, pulse rate) | Screening, up to 20 days after drug administration
Number of patients with abnormal changes in laboratory parameters | Screening, up to 20 days after drug administration
Number of patients with adverse events | up to 41 days
Number of patients with abnormal changes in 12-lead electrocardiogram (ECG) | Screening, up to 20 days after drug administration
Assessment of tolerability by investigator on a 4-point scale | up to 20 days after drug administration